CLINICAL TRIAL: NCT00656253
Title: Clinical Trial on the Effectiveness of Herbal Medicinal Mixture in Parkinson Disease
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Collaborators: State Administration of Traditional Chinese Medicine of the People's Republic of China (Other Government)
Responsible Party: Department of Integrative Medicine, Zhongshan hospital, Zhongshan hospital of Fudan University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2006BAI04A11
Record Dates: First submitted 2008-04-07; First posted 2008-04-11 (Estimated); Last update posted 2011-03-22 (Estimated); Status verified 2009-09

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental)
  Interventions: Drug: Herbal Medicinal Mixture (Roucongrong, Heshouwu etc.)
- B (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Herbal Medicinal Mixture (Roucongrong, Heshouwu etc.) — 12 months period of Herbal Medicinal Mixture per day plus 1 month wash-out period without herbal medicine
  Arms: A
Drug: Placebo — 12 months period of placebo plus 1 month period without placebo
  Arms: B

SUMMARY:
This study was designed to evaluate the symptomatic effects or potential disease progression slowing down effect of a kind of Herbal Medicinal Mixture in Parkinson's disease (PD) patients. The treatment phase includes 12 months period of Herbal Medicinal Mixture per day or placebo and 1 month wash-out period without herbal medicine and placebo.

DETAILED DESCRIPTION:
This study was designed to evaluate the symptomatic effects or potential disease progression slowing down effect of a kind of Herbal Medicinal Mixture in Parkinson's disease (PD) patients. The treatment phase includes 12 months period of Herbal Medicinal Mixture per day or placebo and 1 month wash-out period without herbal medicine and placebo.

The design of the study was a prospective, randomized, multicenter, double-blind placebo-controlled protocol. The intervention includes Herbal Medicinal Mixture Bid or matched placebo for 12 months plus 1 month wash-out period.

Participating study centers include Neurological University Outpatient Clinics and Neurological Departments of Community-based Hospitals experienced with PD patients.

The primary outcome measure was the combined Unified Parkinson's Disease Rating Scale (UPDRS).

The hypothesis of this study was that Herbal Medicinal Mixture improves the overall wellbeing of PD patients and thus may leads to an improvement of parkinsonian symptoms in PD patients.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease according to the UK Brain Bank criteria
* Hoehn & Yahr stadium Ⅰ～Ⅲ
* Age over 50 years
* Taking only levodopa and/or dopamine agonists when recruiting
* Consistent with the liver kidney deficiency type by Traditional Chinese Medicine (TCM) standard
* Patients voluntarily take part in this study and signed the informed consent

Exclusion Criteria:

* Modified Hoehn-Yahr scale are higher than 4
* Had other serious illness such as liver/kidney failure, serious infection etc
* Allergic to the study drug
* Had been participated in other clinical trials during the last 3 months prior to study inclusion.
* Taking Coenzyme Q10, MAO-B inhibitors, or vitamin E, all of which might improve the symptom or slowdown the progression of PD.
* Taking herbal medicine that can nourish the liver and kidney by TCM standard.
* Had serious mental disorder and could not describe his/her symptom.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2008-08; Primary Completion 2010-09 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Levodopa equivalent dose(LED) per day | 13 months
  daily levodopa dose taken by PD patients to control their symptoms.

SECONDARY OUTCOMES:
Unified Parkinson's Disease Rating Scale (UPDRS) | 13 months
Hoehn & Yahr scale | 13 months
Schwab & England score | 13 months
The liver kidney deficiency scale score by Traditional Chinese Medicine standard | 13 months
Parkinson disease sleep scale (PDSS) | 13 months
Assessment of autonomic dysfunction in Parkinson disease (SCOPA-AUT) | 13 months
Changes in laboratory indexes as safety assessment, including red blood cell(RBC), white blood cell(WBC), platelet(PLT), alanine transaminase (ALT), aspartate transaminase (AST), blood urea nitrogen (BUN), creatinine(Cr) in blood samples, ect. | 12 months

CONTACTS AND LOCATIONS:
Locations (10):
- China (10):
  - Department of Neurology, Xuanwu hospital, Capital University of Medical Sciences, Beijing, Beijing Municipality
  - Department of Neurology, Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Department of Integrative Medicine, Zhongshan hospital, Fudan University, Shanghai, Shanghai Municipality
  - Department of Nuerology, Longhua Hospital Affiliated to Shanghai University of Traditional Chinese Medicine, Shanghai, Shanghai Municipality
  - Tongji Hospital of Tongji University, Shanghai, Shanghai Municipality
  - Shanghai Chinese Medical Hospital, Shanghai, Shanghai Municipality
  - Department of Nuerology, Xinhua Hospital, Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - The Sixth People's Hospital, Shanghai Jiaotong University, Shanghai, Shanghai Municipality
  - Department of Neurology, Yueyang Hospital of Traditional Chinese and Western Medicine, Shanghai University of Traditional Chinese Medicine, Shanghai, Shanghai Municipality
  - Department of Neurology, The second people's hospital of Wenzhou, Wenzhou, Zhejiang